CLINICAL TRIAL: NCT00890253
Title: A Therapeutic Exploratory Study to Determine the Efficacy and Safety of Calcineurin-Inhibitor-Free De-novo Immunosuppression After Liver Transplantation
Brief Title: Safety Study of Calcineurin-Inhibitor-Free Immunosuppression After Liver Transplantation
Acronym: CILT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armin Goralczyk (Other)
Responsible Party: Sponsor-Investigator, Armin Goralczyk, Dr., University Medical Center Goettingen
Organization: University Medical Center Goettingen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CILT08
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2010-01

CONDITIONS: Liver Transplantation; Chronic Renal Insufficiency
Keywords: Renal impairment; Liver transplantation; Chronic Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Basiliximab; Mycophenolic Acid; Everolimus; Prednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CNI-free Immunosuppression (Experimental): Immunosuppression after OLT including basiliximab, enteric-coated mycophenolate sodium (EC-MPS), and everolimus.
  Interventions: Drug: Basiliximab (Simulect); Drug: Myfortic; Drug: everolimus; Drug: Prednisolone

INTERVENTIONS:
Drug: Basiliximab (Simulect) — 20 mg basiliximab (Simulect) iv on day 0 and 4 after OLT
  Other Names: Basiliximab: Simulect
Drug: Myfortic — 1080 mg q12 EC-MPS (Myfortic) po starting within 24h after OLT
  Other Names: Enteric-coated mycophenolate sodium: EC-MPS, Myfortic
Drug: everolimus — 1 mg q12 everolimus (Certican) po starting on 10th post-operative day
  Other Names: Certican
Drug: Prednisolone — Prednisolone 1mg per kg body weight starting within 24 hours after transplantation. Then q24 but with reduction by 5 mg every 48 hours until maintenance dose of 7.5 mg
  Other Names: Prednisone

SUMMARY:
A prospective, non-randomized two stage monocentric phase II clinical trial to evaluate a de-novo calcineurin-inhibitor (CNI)-free immunosuppressive regimen based on induction therapy with anti-CD25 monoclonal anti-body (basiliximab), mycophenolic acid (MPA), and mammalian target of rapamycin (mTOR) - inhibition with everolimus to determine its safety and to investigate the preliminary efficacy in patients with impaired renal function at the time-point of liver transplantation (OLT) with regards to the incidence of steroid resistant acute rejection within the first 30 days after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing primary liver transplantation.
2. Patients older than 18 years.
3. Patients with a hepatorenal syndrome.
4. Female patients of childbearing potential willing to perform a highly effective contraception during the study and 12 weeks after conclusion of study participation.
5. eGFR < 50 ml/min at the time point of transplantation.
6. Serum creatinine levels > 1.5 mg/dL at the time-point of transplantation.

Exclusion Criteria:

1. Patients with pre-transplant renal replacement therapy > 14 days.
2. Patients with a reason for renal impairment other than a hepatorenal syndrome.
3. Patients with a known hypersensitivity to mTOR-inhibitors.
4. Patients with a known hypersensitivity to mycophenolate acid.
5. Patients with a known hypersensitivity to anti CD 25-monoclonal antibodies.
6. Patients with platelets < 50.000/nl prior to initiation of therapy with mTOR inhibition.
7. Patients with triglycerides > 350 mg/dl and cholesterol > 300 mg/dl refractory to optimal medical treatment prior to initiation of therapy with mTOR inhibition.
8. Severe systemic infections and wound-healing disturbances.
9. Multiple organ graft recipients.
10. Patients with signs of a hepatic artery stenosis directly prior to initiation of therapy with everolimus.
11. Pregnant women will not be included in the study.
12. Patients with a psychological, familial, sociologic or geographic condition potentially hampering compliance with the study protocol and follow-up schedule.
13. Patients under guardianship (e.g., individuals who are not able to freely give their informed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Steroid resistant rejection | 30 days

SECONDARY OUTCOMES:
Steroid resistant rejection | 1 year
Liver function | 1 year
Calculated glomerular filtration rate | 1 year
Patient survival | 1 year
Number of days on renal replacement therapy | 1 year
Graft survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aiman Obed, PD Dr., Study Director — University Medical Center Goettingen; Armin D Goralczyk, Dr., Principal Investigator — University Medical Center Goettingen
Locations (1):
- University Medical Center Goettingen, Göttingen, Germany

REFERENCES:
- [Derived] Goralczyk AD, Schnitzbauer A, Tsui TY, Ramadori G, Lorf T, Obed A. A therapeutic exploratory study to determine the efficacy and safety of calcineurin-inhibitor-free de-novo immunosuppression after liver transplantation: CILT. BMC Surg. 2010 Apr 9;10:15. doi: 10.1186/1471-2482-10-15. PMID 20380712